CLINICAL TRIAL: NCT04126525
Title: NeoAdjuvant Trastuzumab/ Pyrotinib Plus Weekly Paclitaxel/Cisplatin in HER2-positive Locally Advanced Breast Cancer Patients
Brief Title: Neoadjuvant Study of Pyrotinib in HER-2 Positive Breast Cancer
Acronym: NeoATP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2019-023
Record Dates: First submitted 2019-10-06; First posted 2019-10-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Female
Keywords: neoadjuvant; pyrotinib; trastuzumab; paclitaxel; cisplatin
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant pyrotinib (Experimental): pyrotinib 400mg qd trastuzumab 4mg/kg loading dose, then 2mg/kg qw palitaxel 80mg/m^2, d1, 8, 15, 22 cisplatin 25mg/m^2, d1, 8, 15 every 28 days
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — dual HER2 blockade in the neoadjuvant setting

SUMMARY:
This is a prospective, open label study to evaluate the efficacy and safety of neoadjuvant pyrotinib in early breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female, Aged ≥18 and ≤70 years
* Histologically confirmed invasive HER2 positive breast cancer, early disease(Stage ⅡA-Ⅲ)
* Subjects with at least one evaluable lesion
* ECOG 0-1
* Adequate organ function

Exclusion Criteria:

* Metastatic disease (Stage IV)
* Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption
* Treated or treating with T-DM1, lapatinib and neratinib before study entry
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation
* Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test. Female patients of childbearing age that are reluctant to take effective contraceptive measures throughout the trial period
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
pCR | 1-2 weeks after surgery
  pathological complete response

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Lu, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yin W, Wang Y, Wu Z, Ye Y, Zhou L, Xu S, Lin Y, Du Y, Yan T, Yang F, Zhang J, Liu Q, Lu J. Neoadjuvant Trastuzumab and Pyrotinib for Locally Advanced HER2-Positive Breast Cancer (NeoATP): Primary Analysis of a Phase II Study. Clin Cancer Res. 2022 Sep 1;28(17):3677-3685. doi: 10.1158/1078-0432.CCR-22-0446. PMID 35713517